CLINICAL TRIAL: NCT06993090
Title: Efficacy of the Dorsal Application of Kinesio Tape on Esport Gamers
Brief Title: Efficacy of Dorsal Kinesio Tape Application for Carpal Tunnel Syndrome in Esports Gamers: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNLV-2024-458
Record Dates: First submitted 2025-04-23; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel; Carpal Tunnel Syndrome (CTS)
Keywords: carpal tunnel; carpal tunnel syndrome; gamers; PC gamers; Esports; First person shooter; Kinesiotape
MeSH Terms: conditions — Median Neuropathy; Carpal Tunnel Syndrome | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: The intervention group will receive Kinesio Tape application to the dorsal side of the wrist while the control group will have Kinesio Tape applied to the spine of the Scapula
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Kinesio Tape on Dorsal Wrist (Experimental): Participants in this group will receive Kinesio Tape applied to the dorsal side of the wrist. This application is intended to provide support and potentially reduce carpal tunnel-like symptoms while assessing its impact on gaming performance.
  Interventions: Device: Kinesio Tape
- Kinesio Tape on Scapular Spine (Sham Comparator): Participants in this group will receive Kinesio Tape applied to the scapular spine on the opposite side of their dominant hand. This serves as a control condition to account for the effects of Kinesio Tape placement while ensuring that participants remain blinded to their group assignment.
  Interventions: Device: Kinesio Tape

INTERVENTIONS:
Device: Kinesio Tape — A thin, flexible, and elastic therapeutic tape intended for skin application to provide support for muscles and joints. This tape may help decrease pain, swelling, and inflammation while permitting movement. It is commonly utilized to enhance athletic performance and facilitate injury recovery. The tape functions by elevating the skin, which can enhance blood and lymph circulation, and is believed to engage the nervous system through proprioceptive feedback.

SUMMARY:
This clinical trial investigates the effectiveness of Kinesio Tape (KT) in alleviating carpal tunnel-like symptoms and enhancing gaming performance among young adult PC gamers. The study aims to address two primary questions:

Does Kinesio Tape reduce wrist pain in adult PC gamers experiencing carpal tunnel-like symptoms?

Does Kinesio Tape improve gaming performance in this population?

Researchers will compare the effects of KT applied to the wrist versus the scapular spine to determine if wrist application provides greater pain relief and performance benefits.

Participants will undergo:

Screening & Consent (Up to 30 minutes via Zoom): Informed consent and a Phalen's test to assess carpal tunnel-like symptoms.

Baseline (Day 0, 75 minutes): Completion of a demographic survey, 15 minutes of gaming on Kovaaks FPS Aim Trainer, KT application, 15 minutes of post-application gaming, and surveys (Boston Carpal Tunnel Syndrome Severity [BCSS] and KT feedback).

Days 1 & 2 (15 minutes each): KT removal and reapplication, followed by BCSS and KT feedback surveys.

Day 3 (75 minutes): Repeat gaming tests, KT application, and completion of BCSS and KT feedback surveys, mirroring Day 0 procedures.

Total Time Commitment: Approximately 210 minutes (3.5 hours) over four sessions.

ELIGIBILITY:
* Over 18 years of age
* Test positive for Phalen's screening
* Experience any carpal tunnel-like symptoms
* Self Identified PC gamer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Carpal Tunnel-Like Symptom Severity (Boston Carpal Tunnel Questionnaire - Symptom Severity Scale) | Administered at the end of each session on Day 0 (baseline), Day 1, Day 2, and Day 3 (post-intervention). Sessions were held every other day over an 8-day period.
  This outcome measures the severity and frequency of carpal tunnel-like symptoms, including pain, numbness, tingling, and weakness in the hand, wrist, and forearm. Symptom severity was assessed using the Boston Carpal Tunnel Questionnaire - Symptom Severity Scale (BCTQ-SSS), a validated self-report measure. The BCTQ-SSS uses a 5-point Likert scale where 1 indicates no symptoms and 5 indicates very severe symptoms. Participants rated their symptoms at the end of each session to monitor changes across the intervention period. Higher scores reflect greater symptom burden. This measure was used to evaluate whether kinesiotape application reduced the severity of symptoms commonly associated with repetitive strain injuries in esports players.
Esports Gaming Performance (Kovaaks Aim Trainer) | Day 0 (baseline session) and Day 3 (post-intervention session). In both sessions, performance was measured twice - once before and once after kinesiotape application. Study sessions were conducted every other day over an 8-day period.
  Gaming performance was assessed using Kovaaks Aim Trainer, a validated simulation platform designed to measure key motor skills essential to first-person shooter (FPS) gameplay, including speed, accuracy, reaction time, and total task score. Participants completed two structured testing sessions-on Day 0 (baseline) and Day 3 (post-intervention)-each consisting of 15-minute gaming tasks both before and after kinesiotape application. The selected simulations targeted core esports competencies such as tracking (sustained aim on moving targets), flicking (rapid target shifts), and strafing (aiming while moving), which reflect real-world gaming demands. Performance data, including accuracy percentage and total score, were automatically recorded by the Kovaaks software and later averaged across trials to reduce variability. The purpose of this measure was to evaluate whether kinesiotape-applied to either the dorsal wrist or scapular spine, depending on group assignmet

OTHER OUTCOMES:
Perceived Effects of Kinesiotape (Custom Feedback Questionnaire and Thematic Analysis) | Collected at the end of each session on Day 0 (baseline), Day 1, Day 2, and Day 3 (post-intervention). Sessions were held every other day over an 8-day period.
  This outcome captures participants' subjective perceptions of kinesiotape following each application session. A custom-designed feedback questionnaire was used to collect both quantitative Likert-scale ratings and open-ended qualitative responses. Quantitative items assessed sensations such as tightness, itchiness, and comfort, as well as perceived changes in speed, agility, and overall performance during gameplay. Open-ended responses allowed participants to describe in their own words how the tape influenced their motor control, posture, comfort, and focus. Thematic analysis was used to extract and categorize recurring themes across responses, including enhanced motor precision, ergonomic awareness, sensory experience, and psychological impact. Participants frequently reported improved wrist stability, increased awareness of movement patterns, postural corrections, and heightened confidence in gameplay execution. The integration of qualitative and quantitative feedback provided a ri

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Musculoskeletal Lab, Las Vegas, Nevada
  - Black Fire Innovation, Las Vegas, Nevada
  - Tonopah Residence Complex, Las Vegas, Nevada